CLINICAL TRIAL: NCT07193316
Title: Real Life Safety and Efficacy of Atezolizumab-Bevacizumab Versus Tyrosin Kinase Inhibitors in Patients With Liver Cirrhosis
Brief Title: Safety and Efficacy of Atezolizumab-Bevacizumab Versus Tyrosin Kinase Inhibitors in Patients With Liver Cirrhosis
Acronym: SEEK
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Ponziani Francesca Romana, Dr, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5890
Record Dates: First submitted 2024-04-05; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis
Keywords: hepatocellular carcinoma; atezolizumab bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients receiving atezolizumab/bevacizumab: 247 patients with advanced HCC that received Atezolizumab Bevacizumab
  Interventions: Other: no intervention
- patients receiving tyrosine kinase inhibitors: 494 patients treated with Sorafenib or Lenvatinib per advanced HCC
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Following the results of the randomized clinical trial IMbrave150, the combination of Atezolizumab with Bevacizumab became the first line regimen for patients with advanced hepatocellular carcinoma and it was approved by the FDA and the EMA. Despite these results, real life data on safety and efficacy of this therapy are still lacking. The unmet needs currently observed are: the safety and efficacy in patients with mild liver decompensation (Child Pugh B class) detected before or during treatment start and the role of liver decompensation compared to TKIs therapy. Liver decompensation is not necessary associated with tumor progression and it may occur in patients with liver cirrhosis. Its prognostic role is not known. in this multicentric observational study the Authors enrolled patients with liver cirrhosis and advanced hepatocellular carcinoma treated with Atezolizumab/Bevacizumab to analyse efficacy, safety compared to a retrospectively collected matched cohort of patients treated with TKIs. Moreover They evaluated the safety and efficacy of Atezolizumab/Bevacizumab according to liver function (detected as Child Pugh score and Albumin-Bilirubin grade), underlying etiology of liver disease, presence or absence of portal hypertension and finally presence or absence of liver decompensation. Furthermore, the Authors evaluated its prognostic role on overall survival and time to progression.

DETAILED DESCRIPTION:
Following the results of the randomized clinical trial IMbrave150, the combination of Atezolizumab with Bevacizumab became the first line regimen for patients with advanced hepatocellular carcinoma and it was approved by the FDA and the EMA. Despite these results, real life data on safety and efficacy of this therapy are still lacking. The unmet needs currently observed are: the safety and efficacy in patients with mild liver decompensation (Child Pugh B class) detected before or during treatment start and the role of liver decompensation compared to TKIs therapy. Liver decompensation is not necessary associated with tumor progression and it may occur in patients with liver cirrhosis. Its prognostic role is not known. in this multicentric observational study the Authors enrolled patients with liver cirrhosis and advanced hepatocellular carcinoma treated with Atezolizumab/Bevacizumab to analyse the safety and efficacy compared to a retrospectively collected matched cohort of patients treated with TKIs. Moreover they evaluated the safety and efficacy of Atezolizumab/Bevacizumab according to liver function (detected as Child Pugh score and Albumin-Bilirubin grade), underlying etiology of liver disease, presence or absence of portal hypertension and finally presence or absence of liver decompensation. Furthermore, they evaluated its prognostic role on overall survival and time to progression.

ELIGIBILITY:
Inclusion Criteria:

patients with liver cirrhosis (Child Pugh A or Child Pugh B) and advanced HCC eligible for systemic therapy

* radiological or histological diagnosis of HCC
* age > 18 years old

Exclusion Criteria:

* age < 18 years old
* patients without HCC or with HCC eligible for curative or locoregional treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with liver cirrhosis (Child Pugh A or Child Pugh B) and advanced HCC eligible for systemic therapy
  * radiological or histological diagnosis of HCC
  * age > 18 years old
  exclusion criteria
  * age < 18 years old
  * patients without HCC or with HCC eligible for curative or locoregional treatments
Sampling Method: Non-Probability Sample
Enrollment: 741 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy and safety of Atezolizumab Bevacizumab in terms of overall survival (OS) compard to TKIs. | 2 years
  efficacy and safety of atezolizumab bevacizumab in terms of overall survival

SECONDARY OUTCOMES:
time under treatment | 2 years
  time from the start of treatment to the end of treatment due to any cause
time to decompensation | 2 years
  time from the start of treatment to occurrence of liver decompensation (ascites, bleeding due to portal hypertension, hyperbilirubinemia, hepatic encephalopathy)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160